CLINICAL TRIAL: NCT06108154
Title: Effectiveness of Breastfeeding Techniques to Improve Latching and Prevention of Nipple-soreness Among Primipara Mothers
Brief Title: Effectiveness of Breastfeeding Techniques to Improve Latching and Prevention of Nipplesoreness
Acronym: RCT WHO LATCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Shazia taj, Principal investigator, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LATCH RCT 2007
Record Dates: First submitted 2023-09-28; First posted 2023-10-30 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: 1 SVD group divided into two sub groups. A) interventional.group and B)control group.2. LSCS group divided into two sub groups A)intervention, B)control group.
  observation compare for final result.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational interventional Arm. (Experimental): Interventional arm received educational supportive breastfeeding and hand on training session on Latch techniques according to UNICEF guideline.
  Interventions: Behavioral: Educational breastfeeding traning session
- Control routine hospital care Arm. (No Intervention): Control. No interventions receive hospital routine care

INTERVENTIONS:
Behavioral: Educational breastfeeding traning session — Educational breastfeeding training session base on dialogical, visual attractive and training session on Proper LATCH techniques and breastfeeding positions to prevent from nipplesoreness.
  Other Names: Breastfeeding hands on training session.
  Arms: Educational interventional Arm.

SUMMARY:
There is a significance difference in latch and Nipple-soreness score after intervention in control and interventional. Study population is primiparous mothers.group.interventional group received Breastfeeding supportive educational and training session.control group received hospital routine care.Randomised control trial designed selected. Sample size 60 participants. Latch and nipplesoreness rating scale used for data collection. statistical package of social sciences used for data analysis.outcome utilised in clinical and educative health care system.

DETAILED DESCRIPTION:
Breastfeeding is a natural physiological process but initial critical step on a child s path to a healthy future. Breastfeeding is beneficial to mother, child and society. For this purpose WHO Re-established global breastfeeding culture to promote exclusive breastfeeding (EBF) up-to first 6 months of life 50% by year 2025.Globally Among primiparous 33% mothers experienced breastfeeding problems in first two weeks postpartum. Determinants of premature termination of EBF are nipple soreness, inadequate latch techniques, breast engorgement, and lack of educative supportive system on preventive measures. In Pakistan IMR rate is 55.77% in 2022, major cause is failure to initiate and continuity in breast feeding. Infants get EBF 48% limited to 3 month. One of the significant factor is sore nipples that preeminent by the poor latch contributing 72%, secondary to infants improper sucking. It is hypothesized that ensuring sustain breast feeding by implementing the Planned, educational supportive training sessions, close observation to identify latch related problems and correct them promptly to prevent from nipple soreness, and predict for EBF. The aim of study to determine effectiveness of educational and hand on practice breastfeeding training session to prevent breastfeeding problems that ensure successful breastfeeding journey. Rational of this study is objectively assess the breastfeeding status and take corrective measure before problem become complicated by giving educational breastfeeding training session on preventive basis. However least literature existed on such preventive basis training sessions in countries that have high IMR. The study design will be "Randomized Control Trial." Sample size will comprise of 60 Participants 30 in control and 30 in interventional. Study participants will be selected by non-probability purposive sampling design and allocated in control group and interventional group by Simple Random sampling technique. After signing the informed consent form by participants Demographical data will be elicited. Nipple soreness rating scale and LATCH scoring system will be used to assess the feeding status. Observations will be recorded. SPSS will be used for data analysis and results compare between groups. Independent sample t test will be used to compare the effects of post test score of educational breastfeeding training session. Repeated measure of ANOVA will be used to compare differences between interventional group and control group for weekly follow up if data is normally distributed. A p-value of <0.05 will be considered statistically significant. Outcome utilization of this study, Participants may use independently breastfeeding skills and achieve sustain breastfeeding process. Health care Administrator may make a policy to implement LATCH charting system, (like APGAR score). LATCH scoring system may include in nursing and medical education. Limitations of this study may use limited sample size and lack of follow-ups of infant up-to 6 months. More studies may need to confirm the findings for long term benefits of such training session

ELIGIBILITY:
Inclusion Criteria:

* primiparous mothers in early postpartum with healthy infant outcomes.

Exclusion Criteria:

* Sick mothers.
* Mother with anomaly infants.
* Mothers with contraindication for breastfeeding.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Primiparous mothers.
Enrollment: 100 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
Demographical data, infant Latch on breast. | One month
  Demographical data consisting of socio-demographic characteristics of participants
  1: LATCH scoring system. A systematic breastfeeding assessment, diagnostic and evaluating tool for individual breastfeeding sessions. The tool assigns a numerical score, 0, 1, 2, and includes five key elements of breastfeeding.LATCH: 1. L for infant's ability to latch onto the breast, 2 .A for the presence of audible swallowing of the infant at the breast, 3.T for mother's nipple type, 4.C for mother's sense of comfort,5.H for holding.The total score range from 0 to 10; higher score, the more chances of successful effective breastfeeding. A LATCH score of 0-3 is regarded as poor, 4-7 as moderate/fair, and 8-10 as good/well, during early postpartum. The mothers observed for breastfeeding LATCH by 5-10 minute.

SECONDARY OUTCOMES:
Nipplesoreness | One month
  The nipple soreness rating scale used to determine the pain severity and fissure/cracks on nipples during breastfeeding, 0 = No pain, no tenderness, normal in colour (normal findings), 4 = severe pain, nipple cracked. (Nipple soreness score from 1 to 4 are considered incidence of nipple soreness).

CONTACTS AND LOCATIONS:
Overall Officials: Shazia Taj, Principal Investigator — PG student
Locations (1):
- University of health sciences lahore, Lahore, Punjab Province, Pakistan